CLINICAL TRIAL: NCT03371329
Title: Safety and Feasibility of Mesenchymal Stem Cells Therapy in Patients With Recent Intracerebral Hemorrhage
Brief Title: Mesenchymal Stem Cells Therapy in Patients With Recent Intracerebral Hemorrhage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Abba C. Zubair, M.D., Ph.D., medical Director, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-003524
Record Dates: First submitted 2017-11-03; First posted 2017-12-13 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Hemorrhagic Stroke; Intracerebral Hemorrhage
Keywords: mesenchymal stem cell; stroke; intracerebral hemorrhage; cell therapy
MeSH Terms: conditions — Hemorrhagic Stroke; Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 MSC dose .5 x 10^6/kg IV (Experimental): Intravenous infusion of MSC (mesenchymal stem cell) dose .5 x 10^6/kg for 3 participants.
  Interventions: Biological: MSC
- Group 2 MSC dose 1 x 10^6/kg IV (Experimental): Intravenous infusion of MSC (mesenchymal stem cell) dose 1 x 10^6/kg for next 3 participants.
  Interventions: Biological: MSC
- Group 3 MSC dose 2 x 10^6/kg IV (Experimental): Intravenous infusion of MSC (mesenchymal stem cell) dose 2 x 10^6/kg for next 3 participants.
  Interventions: Biological: MSC
- Group 4 MSC dose 0.5 x 10^6/kg I (Experimental): Intraventricular infusion of MSC (mesenchymal stem cell) dose .5 x 10^6/kg for final 3 participants.
  Interventions: Biological: MSC

INTERVENTIONS:
Biological: MSC — bone marrow derived cultured MSC (mesenchymal stem cell)

SUMMARY:
The overall goal of this study is to develop mesenchymal stem cell therapy for treatment of acute spontaneous hemorrhagic stroke.

DETAILED DESCRIPTION:
The overall clinical development strategy of this project is to conduct this Phase I dose escalation study entitled "A Pilot Study to Evaluate the Safety and Feasibility of Mesenchymal Stem Cells Therapy in Patients with Recent Intracerebral Hemorrhage". This study will be performed under this current IND application and will be limited to the proposed 12 subjects (3 IV and 1 IT dose groups).

In this application the investigators are proposing to evaluate safety and feasibility of allogeneic, bone marrow (BM) derived mesenchymal stem cells (MSC) to induce neuroregeneration, improve neurological function and alleviate inflammation.

ELIGIBILITY:
* Age range: 18 years or older
* Gender: Male or female
* Acute spontaneous supratentorial ICH documented by head CT with ICH Score between 2 - 4 inclusive
* Stable ICH hematoma volume 60mL or less as measured by ABC2 method by 24-72hrs
* Ability to be enrolled within 72 hours of onset of stroke symptoms
* Ability to provide written personal or surrogate consent. Only subjects who have signed the ICF will be enrolled into the study. The ICF will include elements required by Mayo IRB and FDA in US 21CFR50.
* Subject must have adequate renal function; creatinine <1.5g/dl.
* Subject must be available for all specified assessments at the study site through the completion of the study.
* Subject must provide written ICF and authorization for use of and disclosure of PHI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | 1 year
  Number of adverse events at each Mesenchymal Stem Cell (MSC) dose and following infusions up to one year.

SECONDARY OUTCOMES:
Changes in neurological function test | Pre infusion and post-infusion days 1, 2, 3, 7, 30, 90, 180
  The NIH Stroke Scale will be used to assess stroke-related neurologic deficits. A trained observer rates the patient's ability to perform tasks and answer questions. Ratings for each item are scored with 3 to 5 grades with 0 as normal.

CONTACTS AND LOCATIONS:
Overall Officials: Abba C Zubair, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials